CLINICAL TRIAL: NCT04981769
Title: POC SARS-CoV-2 Diagnostic PCR Device Comparison to FDA Approved Reference PCR Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anavasi Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: 003
Record Dates: First submitted 2021-07-27; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients presenting to clinical sites for Covid-19 testing who are 2 years of age or older.
  Interventions: Diagnostic Test: Covid-19 test

INTERVENTIONS:
Diagnostic Test: Covid-19 test — PCR Covid-19 test

SUMMARY:
Study will assess sensitivity and specificity of AnavasiDx POC PCR device for detection of Covid-19 in patients presenting for testing a clinical sites.

DETAILED DESCRIPTION:
Study will assess sensitivity and specificity of AnavasiDx POC PCR device for detection of Covid-19 in patients presenting for testing a clinical sites using a national laboratory PCR Covid-19 test as reference. This study is following FDA EUA molecular test approval criteria. Study will be conducted in 3 or more geographically diverse clinical sites.

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting to clinical site for Covid-19 testing. Completion of signed written informed consent process.

Exclusion Criteria:

* Inability to complete signed written informed consent process. Younger than 2 years of age. Any contraindication to Covid-19 swab testing

Ages: 2 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible subjects presenting to clinical site for Covid-19 testing
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-02 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Covid-19 PCR test result | 90 minutes
  Molecular Covid-19 testing

IPD SHARING:
Plan to Share IPD: No